CLINICAL TRIAL: NCT05263141
Title: Single-center, Prospective, Non-Randomized Control Clinical Trial of Retro-Auricular Single-Site Endoscopic Versus Open Surgery in Patients With Early Stage Papillary Thyroid Carcinoma
Brief Title: Retro-Auricular Single-Site Endoscopic to Papillary Thyroid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ouyang Dian, Clinical Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2022-012-02
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: Papillary Thyroid Carcinoma; Thyroidectomy; Laparoscopy; Retroauricular approach; Single-site
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RASSET group (Experimental): Patients in the retro-auricular single-site endoscopic thyroidectomy (RASSET) group will receive endoscopic thyroid lobectomy and central lymph node dissection.
  Interventions: Procedure: retro-auricular single-site endoscopic thyroidectomy
- traditional open thyroid lobectomy group (Active Comparator): Patients in the traditional open thyroid lobectomy group will receive thyroid lobectomy and central lymph node dissection.
  Interventions: Procedure: traditional open surgery thyroidectomy

INTERVENTIONS:
Procedure: retro-auricular single-site endoscopic thyroidectomy — The strap muscles and the sternocleidomastoid muscle were separated. Upper parathyroid and lower parathyroid glands were identified and preserved. The recurrent laryngeal nerve (RLN) was identified，A lobe of thyroid specimen and central lymph nodes were dissected.
  Other Names: RASSET
  Arms: RASSET group
Procedure: traditional open surgery thyroidectomy — The strap muscles were separated in the midline to expose the thyroid gland. Upper parathyroid and lower parathyroid glands were identified and preserved. The recurrent laryngeal nerve (RLN) was identified， a lobe of thyroid specimen and central lymph nodes were dissected.
  Arms: traditional open thyroid lobectomy group

SUMMARY:
The goal of this non randomized control clinical research study is to compare the cosmetic outcomes and efficiacy of retro-auricular single-site endoscopic thyroid lobectomy and central lymph node dissection against conventional resection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, no gender restrictions.
2. Fine-needle aspiration cytology(FNA) confirmed papillary thyroid carcinoma(PTC).
3. Early stage PTC (stage T1N0M0).
4. Preoperative ultrasonography showed unilateral glandular lobe malignant tumor and the largest diameter was not more than 2cm, without cervical lymph node metastasis and extensive metastasis.
5. Patients undergoing thyroid lobectomy and central lymph node dissection.
6. Patients who have signed an approved Informed Consent.

Exclusion Criteria:

1. Patients who do not accept case data collection for various reasons.
2. The clinical data unfit this study (at the discretion of the investigator).
3. Patients who have undergone neck surgery or radiotherapy before this trail.
4. Patients who have uncontrolled hyperthyroidism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
postoperative cosmetic satisfaction scores | 3 months from surgery
  The cosmetic satisfaction score(CSS) was defined as the sum of the scores on questions about the scar. Q1 and Q2 was using a verbal response scale from 1 to 5 (corresponding to decreasing satisfaction). The other four questions, each on a scale of 0 to 3 (again of decreasing satisfaction).

SECONDARY OUTCOMES:
postoperative Vancouver Scar Scale | 3 months from surgery
  The Vancouver Scar Scale(VSS) is used for scar assessment. It has six domains: vascularity, pigmentation, pliability, height, pain and itchiness. The maximum score for the sum of the domain scores is 18, which corresponds to the worst scar, while 0 indicates normal skin.
postoperative Vancouver Scar Scale | 1 month from surgery
  The Vancouver Scar Scale(VSS) is used for scar assessment. It has six domains: vascularity, pigmentation, pliability, height, pain and itchiness. The maximum score for the sum of the domain scores is 18, which corresponds to the worst scar, while 0 indicates normal skin.
Intra-operative, peri-operative, post-operative clinicopathologic characteristics | 1 week from surgery
  Baseline clinicopathologic characteristics of patients
postoperative cosmetic satisfaction scores | 1 month from surgery
  The cosmetic satisfaction score(CSS) was defined as the sum of the scores on questions about the scar. Q1 and Q2 was using a verbal response scale from 1 to 5 (corresponding to decreasing satisfaction). The other four questions, each on a scale of 0 to 3 (again of decreasing satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Dian Ouyang, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anuwong A, Ketwong K, Jitpratoom P, Sasanakietkul T, Duh QY. Safety and Outcomes of the Transoral Endoscopic Thyroidectomy Vestibular Approach. JAMA Surg. 2018 Jan 1;153(1):21-27. doi: 10.1001/jamasurg.2017.3366. PMID 28877292
- [Background] Lee DW, Ko SH, Song CM, Ji YB, Kim JK, Tae K. Comparison of postoperative cosmesis in transaxillary, postauricular facelift, and conventional transcervical thyroidectomy. Surg Endosc. 2020 Aug;34(8):3388-3397. doi: 10.1007/s00464-019-07113-1. Epub 2019 Sep 12. PMID 31515625
- [Background] Dong F, Ao Y, Li MT, Zhan ZR, Lin YQ, Tan QJ, Li H, Yang AK, Ouyang D. [A comparative study between retro-auricular single-site endoscopic thyroidectomy and transoral endoscopic thyroidectomy vestibular approach: a single-center retrospective analysis]. Zhonghua Wai Ke Za Zhi. 2021 Nov 1;59(11):891-896. doi: 10.3760/cma.j.cn112139-20210903-00420. Chinese. PMID 34743449
- [Background] Schardey HM, Schopf S, Kammal M, Barone M, Rudert W, Hernandez-Richter T, Portl S. Invisible scar endoscopic thyroidectomy by the dorsal approach: experimental development of a new technique with human cadavers and preliminary clinical results. Surg Endosc. 2008 Apr;22(4):813-20. doi: 10.1007/s00464-008-9761-y. Epub 2008 Feb 23. PMID 18297357
- [Background] Berber E, Bernet V, Fahey TJ 3rd, Kebebew E, Shaha A, Stack BC Jr, Stang M, Steward DL, Terris DJ; American Thyroid Association Surgical Affairs Committee. American Thyroid Association Statement on Remote-Access Thyroid Surgery. Thyroid. 2016 Mar;26(3):331-7. doi: 10.1089/thy.2015.0407. PMID 26858014
- [Background] Russell JO, Razavi CR, Al Khadem MG, Lopez M, Saraf S, Prescott JD, Starmer HM, Richmon JD, Tufano RP. Anterior cervical incision-sparing thyroidectomy: Comparing retroauricular and transoral approaches. Laryngoscope Investig Otolaryngol. 2018 Sep 24;3(5):409-414. doi: 10.1002/lio2.200. eCollection 2018 Oct. PMID 30410996
- [Background] Nguyen HX, Nguyen HX, Nguyen HV, Nguyen LT, Nguyen TTP, Le QV. Transoral Endoscopic Thyroidectomy by Vestibular Approach with Central Lymph Node Dissection for Thyroid Microcarcinoma. J Laparoendosc Adv Surg Tech A. 2021 Apr;31(4):410-415. doi: 10.1089/lap.2020.0411. Epub 2020 Jul 17. PMID 32706603
- [Background] Nakajo A, Arima H, Hirata M, Mizoguchi T, Kijima Y, Mori S, Ishigami S, Ueno S, Yoshinaka H, Natsugoe S. Trans-Oral Video-Assisted Neck Surgery (TOVANS). A new transoral technique of endoscopic thyroidectomy with gasless premandible approach. Surg Endosc. 2013 Apr;27(4):1105-10. doi: 10.1007/s00464-012-2588-6. Epub 2012 Nov 21. PMID 23179070
- [Background] Duek I, Duek OS, Fliss DM. Minimally Invasive Approaches for Thyroid Surgery-Pitfalls and Promises. Curr Oncol Rep. 2020 Jun 29;22(8):77. doi: 10.1007/s11912-020-00939-2. PMID 32601931
- [Background] Chung EJ, Park MW, Cho JG, Baek SK, Kwon SY, Woo JS, Jung KY. A prospective 1-year comparative study of endoscopic thyroidectomy via a retroauricular approach versus conventional open thyroidectomy at a single institution. Ann Surg Oncol. 2015 Sep;22(9):3014-21. doi: 10.1245/s10434-014-4361-7. Epub 2015 Jan 21. PMID 25605517
- [Background] Schardey HM, Barone M, Portl S, von Ahnen M, von Ahnen T, Schopf S. Invisible scar endoscopic dorsal approach thyroidectomy: a clinical feasibility study. World J Surg. 2010 Dec;34(12):2997-3006. doi: 10.1007/s00268-010-0769-9. PMID 20835708

DOCUMENTS (1):
  • Study Protocol (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT05263141/Prot_000.pdf